CLINICAL TRIAL: NCT00499291
Title: Pharmacokinetic, Pharmacodynamic and Pharmacogenetic Study of Nab-Paclitaxel (Nanoparticle Albumin Bound-Paclitaxel) in Patients With Advanced Solid Tumors
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Advanced or Refractory Solid Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000554709; ECOG-E1Y06
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Cancer
Keywords: unspecified adult solid tumor, protocol specific; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent bladder cancer; stage III bladder cancer; stage IV bladder cancer; recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; clear cell sarcoma of the kidney; rhabdoid tumor of the kidney; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; fallopian tube cancer; recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent hypopharyngeal cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent laryngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer; recurrent lip and oral cavity cancer; stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; recurrent oropharyngeal cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer; adult central nervous system germ cell tumor; adult teratoma; ovarian teratoma; testicular teratoma; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Testicular Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Teratoma; Teratoma, Ovarian; Teratoma, Testicular; Sarcoma; Neoplasms, Unknown Primary | interventions — Taxes; Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Procedure: gene expression analysis
Procedure: laboratory biomarker analysis
Procedure: pharmacological study
Procedure: polymerase chain reaction

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This clinical trial is studying how well paclitaxel albumin-stabilized nanoparticle formulation works in treating patients with advanced or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To develop a population pharmacokinetic model for paclitaxel administered as paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel) to a large population of patients with advanced or refractory cancer to characterize the inter-individual pharmacokinetic variability of this agent.

Secondary

* To explore nab-paclitaxel pharmacokinetic parameters in patients with metastatic prostate cancer (castrate), metastatic breast cancer, advanced non-small cell lung cancer and other incurable advanced or refractory tumors amenable to treatment with nab-paclitaxel.
* To explore the association between exposure to total and unbound paclitaxel after administration of nab-paclitaxel and neutropenia.
* To explore the association between the CYP2C8*3 variant and paclitaxel clearance.
* To explore the association between other variants of CYP2C8 and other genes involved in paclitaxel disposition including CYP3A4, CYP3A5, SLCO1B3 (OATP8), and ABCB1 (MDR1) and paclitaxel pharmacokinetic parameters and toxicity after one course of treatment.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel) IV over 30 minutes on days 1, 8, 15, 22, 29, 36, 43, and 50. Treatment may repeat off study every 9 weeks in the absence of disease progression or unacceptable toxicity.

Serial blood samplings are obtained at specified time points during course 1 including baseline and days 1 and 8 of course 1 for pharmacokinetic studies. Samples are also examined for genotype by PCR including variant genotypes in 2C8, CYP3A4, CYP3A5, ABCB1, ABCC2, ABCC10 and OATP1B3 genes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must have an incurable advanced or refractory tumor amenable to treatment with paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel)

  * Per the National Comprehensive Cancer Network, the following cancer sites have been shown to be responsive to taxane therapy:

    * Prostate cancer
    * Breast cancer
    * Non-small cell lung cancer
    * Bladder cancer
    * Head and neck cancer
    * Oral cancer
    * Cervical cancer
    * Ovarian cancer
    * Endometrial cancer
    * Esophageal cancer
    * Gastric cancer
    * Germ cell tumors
    * Tumors of unknown primary
    * Soft tissue sarcomas
    * Small cell lung cancer
    * Testicular cancer
    * Upper genitourinary tract cancers

PATIENT CHARACTERISTICS:

* Patients must have performance status 0-2 by the ECOG scale
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ institutional upper limit of normal (ULN)
* ALT and AST ≤ 2.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN (if bone metastasis is present in the absence of liver metastasis, alkaline phosphatase must be ≤ 5 x ULN)
* Creatinine ≤ 1.5 x ULN
* Patients must not have baseline sensory neuropathy ≥ grade 2
* Women must not be pregnant or breastfeeding
* Negative blood or urine pregnancy test
* Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception

PRIOR CONCURRENT THERAPY:

* Prior treatment is allowed, which may include prior taxane therapy

  * If patient has had prior therapy(ies), s/he must have received last treatment ≥ 28 days prior to registration
* Patients must not be receiving colony stimulating factors (CSFs)

  * Previous CSFs must have been discontinued > 14 days prior to registration
* Patients must not be receiving concomitant treatment with any of the following (prior use is allowed, but must have been discontinued ≥ 28 days prior to registration):

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampicin
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
  * Ketoconazole

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Inter-individual pharmacokinetic variability

SECONDARY OUTCOMES:
Pharmacokinetic parameters
Neutropenia
CYP2C8*3 variant expression
Genetic variance relating to pharmacokinetics and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Study Chair — Albert Einstein College of Medicine